CLINICAL TRIAL: NCT01131117
Title: Fetal Programming of Obesity
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 110889
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Pregnancy
Keywords: healthy; women; pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool, human milk, placenta, cord blood and umbilical cord may be collected from study participants.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women

SUMMARY:
The overall goal of this project is to understand how a mother's health at conception may influence her child's growth and development.

DETAILED DESCRIPTION:
The purpose of this study is to determine how the mother's health prior to or at the beginning of pregnancy may influence her child's growth and development. We plan to: 1) longitudinally and simultaneously assess a true measure of body composition (lean and fat mass) of the offspring, assess body composition of both parents, and obtain dietary intake data of the mother and offspring; 2) determine endocrine and metabolic profiles of the mother at baseline (pre-conception), during pregnancy and at birth (such as insulin, glucose, leptin); 3) determine the energy expenditure and physical activity of the mother and the child; 4) determine gene expression of the placenta and umbilical cord via gene microarray and real time PCR; and 5) focused on appropriate-for-gestational age (AGA) infants (the majority of infants born from normal and overweight mothers).Accordingly, this study will provide much needed comprehensive information on the possible effect of fetal programming on the development of pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 21 years of age or older
* second pregnancy, singleton
* conceived without fertility treatments

Exclusion Criteria:

* Preexisting medical conditions
* Sexually transmitted diseases
* Medical complications during pregnancy
* Medications during pregnancy known to influence fetal growth
* Smoking, alcohol drinking
* Excessive physical activity level which could affect the outcome of interest.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2010-04-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Child body composition | 24 months
  lean and fat mass of the child

SECONDARY OUTCOMES:
Child metabolism | 24 months
  monitor with a metabolic cart
Child development | 24 months
  Monitored from 2wks up to 24 months
Child dietary intake | 24 months
  Food records for each visit will be obtained
Placenta gene expression | 9 months
  via gene microarray and real time PCR
Placenta protein content | 9 months
  via gene microarray and real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, RD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Crimmins MR, Hand M, Samuel H, Bellando J, Sims CR, Andres A, Sobik S. The Impact of Excessive Weight on Breastfeeding Intention, Initiation, and Duration. Breastfeed Med. 2023 Sep;18(9):688-695. doi: 10.1089/bfm.2023.0072. PMID 37729033
- [Derived] Gilley SP, Ruebel ML, Sims C, Zhong Y, Turner D, Lan RS, Pack LM, Piccolo BD, Chintapalli SV, Abraham A, Bode L, Andres A, Shankar K. Associations between maternal obesity and offspring gut microbiome in the first year of life. Pediatr Obes. 2022 Sep;17(9):e12921. doi: 10.1111/ijpo.12921. Epub 2022 Apr 27. PMID 35478493
- [Derived] Kracht CL, Redman LM, Casey PH, Krukowski RA, Andres A. Association between Home Environment in Infancy and Child Movement Behaviors. Child Obes. 2021 Mar;17(2):100-109. doi: 10.1089/chi.2020.0319. Epub 2021 Jan 20. PMID 33471594
- [Derived] Saben JL, Sims CR, Piccolo BD, Andres A. Maternal adiposity alters the human milk metabolome: associations between nonglucose monosaccharides and infant adiposity. Am J Clin Nutr. 2020 Nov 11;112(5):1228-1239. doi: 10.1093/ajcn/nqaa216. PMID 32844207
- [Derived] Sims CR, Lipsmeyer ME, Turner DE, Andres A. Human milk composition differs by maternal BMI in the first 9 months postpartum. Am J Clin Nutr. 2020 Sep 1;112(3):548-557. doi: 10.1093/ajcn/nqaa098. PMID 32401302
- [Derived] Allman BR, Diaz EC, Andres A, Borsheim E. Divergent Changes in Serum Branched-Chain Amino Acid Concentrations and Estimates of Insulin Resistance throughout Gestation in Healthy Women. J Nutr. 2020 Jul 1;150(7):1757-1764. doi: 10.1093/jn/nxaa096. PMID 32275314
- [Derived] Diaz EC, Borsheim E, Shankar K, Cleves MA, Andres A. Prepregnancy Fat Free Mass and Associations to Glucose Metabolism Before and During Pregnancy. J Clin Endocrinol Metab. 2019 May 1;104(5):1394-1403. doi: 10.1210/jc.2018-01381. PMID 30496579
- [Derived] Porter H, West DS, Cleves MA, Saylors ME, Andres A, Krukowski RA. Association Between Household Food Environment and Excessive Gestational Weight Gain. J Womens Health (Larchmt). 2018 Aug;27(8):1064-1070. doi: 10.1089/jwh.2017.6552. Epub 2018 Apr 5. PMID 29620954
- [Derived] Krukowski RA, West DS, DiCarlo M, Cleves MA, Saylors ME, Andres A. Association of Gestational Weight Gain Expectations and Advice on Actual Weight Gain. Obstet Gynecol. 2017 Jan;129(1):76-82. doi: 10.1097/AOG.0000000000001780. PMID 27926649
- [Derived] Krukowski RA, West DS, DiCarlo M, Shankar K, Cleves MA, Saylors ME, Andres A. Are early first trimester weights valid proxies for preconception weight? BMC Pregnancy Childbirth. 2016 Nov 21;16(1):357. doi: 10.1186/s12884-016-1159-6. PMID 27871260
- [Derived] Krukowski RA, West D, DiCarlo M, Shankar K, Cleves MA, Tedford E, Andres A. A Behavioral Intervention to Reduce Excessive Gestational Weight Gain. Matern Child Health J. 2017 Mar;21(3):485-491. doi: 10.1007/s10995-016-2127-5. PMID 27449652